CLINICAL TRIAL: NCT03369483
Title: Evaluation of the Abdominal Pressure Modifications in Patients Undergone to Open Abdominal Surgery and Receiving Continuous Positive Airway Pressure
Brief Title: Abdominal Pressure Assessment Following Open Abdominal Surgery
Acronym: AbdoPress
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Paolo Navalesi, MD, University Magna Graecia
Other Study IDs: 284/2017
Record Dates: First submitted 2017-11-29; First posted 2017-12-12 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Lung Collapse
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CPAP: At the end of the abdominal surgical procedure, mechanical ventilation withdrawal and extubation, patients will receive Continuous Positive Airway Pressure CPAP). CPAP will be be delivered using any commercially available CPAP equipment. CPAP will be started as soon as possible after the end of surgery. The starting airway pressure (PEEP) will be 5 cmH2O. PEEP may be changed at the discretion of the responsible physician. The maximum permissible PEEP during the trial intervention period will be 10 cmH2O. CPAP may be continued after the four-hour trial intervention period has finished, at the discretion of the responsible physician.
  Interventions: Other: Abdominal pressure assessment

INTERVENTIONS:
Other: Abdominal pressure assessment — We will perform measurements of the abdominal pressure an urinary catheter connected with an intra-abdominal pressure device (Uno-Meter ® - Unomedical) in all patients undergoing on open-surgical procedures after mechanical ventilation withdrawal and extubation, 30 minutes and 4 hours after the application of CPAP.

SUMMARY:
During abdominal surgery, the intra abdominal pressure may increase determining lung bibasal atelectasis. The investigators hypothesized that the application of Positive End Expiratory Pressure (PEEP) promptly after extubation through Continuous Positive Airway Pressure (CPAP) would improved gas exchange, especially in those patients with abdominal pressure values close to those applied by CPAP.

The investigators have therefore designed this subset study enrolling patients randomized to receive CPAP in the "Prevention of Respiratory Insufficiency after Surgical Management (PRISM)" Trial in order to ascertain the abdominal pressure in post-surgical patients (abdominal open surgery procedures) enrolled in PRISM trial. In addition they would evaluate the effects of CPAP on abdominal pressure and consequently on arterial blood gas, and whether there is a correlation between PEEP values, abdominal pressure values and arterial blood gas.

One hundred patients included in CPAP group of the PRISM trial will be enrolled in this subset study. The investigators will perform measurements of the abdominal pressure an urinary catheter connected with an intra-abdominal pressure device (Uno-Meter ® - Uno-medical) in all patients undergoing on open-surgical procedures after mechanical ventilation withdrawal and extubation, 30 minutes and 4 hours after the application of CPAP.

DETAILED DESCRIPTION:
Major abdominal surgery is associated with adverse changes in respiratory function.

Anaesthesia can cause reduced vital capacity, hypoxaemia and impaired central respiratory drive, while surgical manipulation can restrict ventilation, damage the respiratory muscles and cause atelectasis. These factors interact with pre-existing respiratory disease and postoperative pain to create a significant risk of pneumonia and respiratory failure, which may result in death. Evidence from one study suggests that the risk of mortality within 30 days of surgery is increased from 1% to 27% in patients with respiratory failure. Usual treatments including supplemental oxygen or respiratory physiotherapy may not always prevent deterioration in respiratory function. Subsequent respiratory failure can lead to endotracheal intubation and mechanical ventilation, which is in turn associated with a range of serious morbidities. Continuous positive airway pressure (CPAP) is a non-invasive method of supporting respiratory function. The patient breathes through a pressurized circuit against a threshold resistor that maintains a pre-set positive airway pressure during both inspiration and expiration. The findings of several trials have demonstrated the efficacy of CPAP as preventative treatment for high-risk patients following abdominal surgery by reducing the incidence postoperative pulmonary complications.

The investigators have hypothesized that the application of Positive End Expiratory Pressure (PEEP) promptly after extubation through CPAP would improved gas exchange, especially in those patients with abdominal pressure values close to those applied by CPAP.

The investigators have therefore designed this subset study enrolling patients randomized to receive CPAP in the "Prevention of Respiratory Insufficiency after Surgical Management (PRISM)" Trial in order to ascertain the abdominal pressure in post-surgical patients (abdominal open surgery procedures) enrolled in PRISM trial. In addition they would evaluate the effects of CPAP on abdominal pressure and consequently on arterial blood gas, and whether there is a correlation between PEEP values, abdominal pressure values and arterial blood gas.

One hundred patients included in CPAP group of the PRISM trial will be enrolled in this subset study. To be included in the PRISM trial, patients are required to be 50 years/old or over and to undergo major, open, intra-peritoneal surgery. Patients are excluded of meeting one or more of the following: 1) inability or refusal to provide informed consent; 2) anticipated requirement for invasive or non-invasive mechanical ventilation or at least four hours after surgery as part of routine care; 3) pregnancy or obstetric surgery; 4) previous enrolment in PRISM trial; 5) participation in a clinical trial of a treatment with a similar biological; 6) mechanism or related primary outcome measure and 7) clinician refusal.

CPAP will be provided for at least four hours, with minimal interruption, started soon after the patient has left the operating room after surgery. Administration of CPAP will only take place under the direct supervision of appropriately trained staff in an adequately equipped clinical area. The monitoring of patients receiving CPAP will be in accordance with local hospital policy or guidelines. Alterations to the administered dose will be recorded along with the reason for this change. Clinicians may only use commercially available CPAP equipment to deliver the intervention. The starting airway pressure should be 5 cmH2O and the maximal permissible airway pressure is 10 cmH2O.

The investigators will perform measurements of the abdominal pressure an urinary catheter connected with an intra-abdominal pressure device (Uno-Meter ® - Uno-medical) in all patients undergoing on open-surgical procedures after mechanical ventilation withdrawal and extubation, 30 minutes and 4 hours after the application of CPAP. Moreover, arterial blood will be sample for gas analysis at every aforementioned time-step.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50 years or over undergoing major, open, intra-peritoneal surgery, randomized to receive Continuous Positive Airway Pressure in the "Prevention of Respiratory Insufficiency after Surgical Management (P.R.I.S.M. TRIAL)"

Exclusion Criteria:

* Inability or refusal to provide informed consent
* Anticipated requirement for invasive or non-invasive mechanical ventilation for at least four hours after surgery as part of routine care
* Pregnancy or obstetric surgery
* Previous enrollment in PRISM trial
* Participation in a clinical trial of a treatment with a similar biological mechanism or related primary outcome measure
* Clinician refusal

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We will observe the aforementioned physiologic parameters in 100 patients randomized to receive CPAP treatment in another international multicenter trial (PRISM trial). Patients will be therefore eligible if 50 years old or higher, undergoing major, open, intra-peritoneal surgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-03-13 (Actual); Primary Completion 2021-03-05 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Abdominal pressure in post-surgical patients (abdominal open surgery procedures) | Within 30 minutes by the end of surgery and mechanical ventilation withdrawn
  Assessment of abdominal pressure through a dedicated device connected to the urinary catheter

SECONDARY OUTCOMES:
Abdominal pressure | After 30 minutes from the application of Continuous Positive Airway Pressure
  Assessment of abdominal pressure through a dedicated device connected to the urinary catheter
Abdominal pressure | After 4 hours from the application of Continuous Positive Airway Pressure
  Assessment of abdominal pressure through a dedicated device connected to the urinary catheter
Arterial blood gases | Within 30 minutes by the end of surgery and mechanical ventilation withdrawn
  Sample of arterial blood for gas analysis
Arterial blood gases | After 30 minutes from the application of Continuous Positive Airway Pressure
  Sample of arterial blood for gas analysis
Arterial blood gases | After 4 hours from the application of Continuous Positive Airway Pressure
  Sample of arterial blood for gas analysis

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Navalesi, MD, Principal Investigator — Magna Graecia University, Catanzaro, Italy
Locations (5):
- Italy (5):
  - Magna Graecia University - University Hospital Mater Domini, Catanzaro
  - Dipartimento di Morfologia, Chirurgia e Medicina Sperimentale, Sezione di Anestesiologia e Terapia Intensiva Universitaria, Università degli studi di Ferrara, Ferrara
  - Department of Anesthesia and Intensive Care, IRCCS Policlinic San Matteo Hospital Foundation , Pavia , Italy, Pavia
  - Anesthesia and Intensive Care Medicine, Sapienza University of Rome, Policlinico Umberto I Hospital, Roma
  - University of Sassari, Sassari

IPD SHARING:
Plan to Share IPD: Undecided